CLINICAL TRIAL: NCT06007690
Title: A Phase 3 Randomized, Masked, Controlled Trial to Evaluate Efficacy and Safety of Belzupacap Sarotalocan (AU-011) Treatment Compared to Sham Control in Subjects With Primary Indeterminate Lesions or Small Choroidal Melanoma
Acronym: CoMpass
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AU-011-301
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Choroidal Melanoma; Indeterminate Lesions; Uveal Melanoma; Ocular Melanoma
Keywords: Uveal Melanoma; Eye Cancer; Ocular Melanoma; Choroidal Melanoma
MeSH Terms: conditions — Uveal Melanoma; Eye Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject, Assessor, and Sponsor masked trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- High dose bel-sar treatment arm & laser application (Experimental): High dose of bel-sar + laser application
  Interventions: Drug: Bel-sar; Device: Suprachoroidal Microinjector; Device: Infrared Laser
- Low dose bel-sar treatment arm & laser application (Experimental): Low dose of bel-sar + laser application
  Interventions: Drug: Bel-sar; Device: Suprachoroidal Microinjector; Device: Infrared Laser
- Sham control arm & sham laser (Sham Comparator): Sham injection + sham laser
  Interventions: Device: Sham Infrared Laser; Device: Sham Microinjector

INTERVENTIONS:
Drug: Bel-sar — Bel-sar via suprachoroidal administration followed by laser application.
  Other Names: AU-011
  Arms: High dose bel-sar treatment arm & laser application; Low dose bel-sar treatment arm & laser application
Device: Suprachoroidal Microinjector — Suprachoroidal injection device
  Other Names: SCS Microinjector
  Arms: High dose bel-sar treatment arm & laser application; Low dose bel-sar treatment arm & laser application
Device: Infrared Laser — Laser application
  Arms: High dose bel-sar treatment arm & laser application; Low dose bel-sar treatment arm & laser application
Device: Sham Infrared Laser — Sham laser application
  Arms: Sham control arm & sham laser
Device: Sham Microinjector — Sham injection device
  Arms: Sham control arm & sham laser

SUMMARY:
The primary objective is to determine the safety and efficacy of belzupacap sarotalocan (bel-sar) compared to sham control in patients with primary indeterminate lesions (IL) or small choroidal melanoma (CM).

DETAILED DESCRIPTION:
This is a randomized, sham-controlled, subject-, assessor-, and Sponsor- masked trial to establish the safety and efficacy of bel-sar treatment via suprachoroidal (SC) administration in subjects with primary IL/CM. Bel-sar treatment incorporates administration of bel-sar drug product using a suprachoroidal space (SCS) microinjector and activation of bel-sar by a laser photoactivation device.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary indeterminate lesion or small choroidal melanoma (IL/CM)
* Have no evidence of metastatic disease confirmed by imaging
* Be treatment naive for IL/CM (subjects who received PDT may be eligible)

Exclusion Criteria:

* Have known contraindications or sensitivities to the study drug or laser
* Active ocular infection or disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Time to reach tumor progression | 65 weeks
  Tumor Progression

SECONDARY OUTCOMES:
Time to composite endpoint | 65 weeks
  Tumor progression or visual acuity failure

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Aura Biosciences
Locations (66):
- United States (35):
  - Retina Consultants of Alabama, Birmingham, Alabama
  - UCSD Shiley Eye Institute, Jacobs Retina Center, La Jolla, California
  - Doris Stein Eye Research Center, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Retina Associates of Florida, PA, Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Tufts Medical Center New England Eye Center, Boston, Massachusetts
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - W.K. Kellogg Eye Center - University of Michigan, Ann Arbor, Michigan
  - Associated Retinal Consultants (ARC) P.C., Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Medicine's Truhlsen Eye Institute, Omaha, Nebraska
  - Columbia University Irving Medical Center, New York, New York
  - Duke Eye Center, Durham, North Carolina
  - Cole Eye Institute, Cleveland, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Consultants of Oklahoma, Oklahoma City, Oklahoma
  - Shields & Shields PC-Wills Eye Institute, Philadelphia, Pennsylvania
  - Retina Consultants of Carolina, Greenville, South Carolina
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Tennessee Retina, PC, Nashville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - UT, Southwestern Medical Center, Dallas, Texas
  - Retina Associates of South Texas, P.A., San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Vitreoretinal Associates of Washington, Bellevue, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Madison, Madison, Wisconsin
- Australia (2):
  - Terrace Eye Centre, Brisbane, Queensland
  - Eye Research Australia, East Melbourne, Victoria
- Austria (2):
  - Medical University Graz, Graz
  - Medizinische Universität Wien, Department of Ophthalmology and Optometry, Vienna
- UZ Leuven, Leuven, Belgium
- Canada (3):
  - Serac Eye and Skin Care Centre, Calgary, Alberta
  - Princess Margaret Eye Tumour Clinic, Toronto, Ontario
  - Centre Hospitalier de l'Universite Laval, Québec, Quebec
- Czechia (3):
  - Fakultni Thomayerova nemocnice, Prague, Krč
  - Fakultni nemocnice Plzen, Pilsen, Plzenský Kraj
  - Ustredni vojenska nemocnice Vojenska fakultni nemocnice Praha, Prague
- Centre Hospitalier Universitaire de Nice, Nice, Cedex 1, France
- Germany (5):
  - Charité - Universitätsmedizin Berlin KöR, Berlin
  - Uniklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Schleswig-Holstein Klinik für Augenheilkunde, Lübeck
  - Klinikum der LMU Muenchen, München
  - Universitätsklinikum Tübingen, Tübingen
- Israel (2):
  - The Chaim Sheba Medical Center, Tel-Hashomer, Central District
  - Hadassah Medical Center, Ein-Karem, Jerusalem, Jerusalem
- Italy (4):
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Nazionale dei Tumori, Fondazione IRCCS, Milan
  - Ospedale Fatebenefratelli e Oftalmico, ASST Fatebenefratelli Sacco, Milan
  - Universita'Cattolica Del Sacro Cuore - UNICATT, Roma
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Erasmus MC, Rotterdam
- Auckland Eye Ltd, Auckland, New Zealand
- Spain (3):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Provincial de Conxo, Santiago de Compostela
  - Hospital Universitario Y Politécnico La Fe, Valencia
- United Kingdom (2):
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Nhs Foundation Trust - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aura Biosciences — http://www.aurabiosciences.com